CLINICAL TRIAL: NCT06667037
Title: Myopia Control Effect of Orthokeratology and 0.01% Atropine Sequential Treatment in Children and Adolescents: A Multicenter Randomized Controlled Trial
Brief Title: Orthokeratology and 0.01% Atropine Sequential Treatment for Myopia Control
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Collaborators: People's Hospital of Guangxi (Unknown); Henan Provincial People's Hospital (Unknown); Tianjin Medical University Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024KYPJ103
Record Dates: First submitted 2024-10-14; First posted 2024-10-31 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Atropine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ortho-k and 0.01% atropine sequential treatment (Experimental): Participants will be treated with ortho-k lenses during the first year, and swiched to recieve 0.01% atropine twice a day in the second year.
  Interventions: Device: Ortho-k lenses; Drug: 0.01% Atropine
- Ortho-k continuous treatment (Active Comparator): Participants will be treated with ortho-k lenses throughout, during the 2-year study period.
  Interventions: Device: Ortho-k lenses

INTERVENTIONS:
Device: Ortho-k lenses — Ortho-k lenses will be administered nightly.
Drug: 0.01% Atropine — 0.01% Atropine will be administrated twice a day with an interval of about 12 hours. Drop into the conjunctival sac and immediately compress the lacrimal sac of the inner canthus for 2-3 minutes.
  Arms: Ortho-k and 0.01% atropine sequential treatment

SUMMARY:
The purpose of this multicenter randomized clinical trial is to evaluate the myopia control effect of orthokeratology and 0.01% atropine sequential treatment in children and adolescents, as compared to continuous treatment with orthokeratology.

DETAILED DESCRIPTION:
Myopia constitutes a major threat to vision health globally for its increasing prevalence and irriversible blinding complications. It is crucial to effectively intervene subjects with progressive myopia to reduce risks of myopic pathologies in later life.

Orthokeratology (ortho-k) is the first-line intervention for myopia control, with an efficacy of slowing axial elongation by 43-63%. However, the efficacy decreases over time. Sequential treatment strategy, which switches myopia control interventions at some intervals, has a potential to increase myopia control efficacy regarding the whole treatment period, compared to applying one intervention throughout. However, there lacks evidence supporting the benefit of this treatment strategy.

The purpose of this study is to evaluate the effectiveness of orthokeratology and 0.01% atropine sequential treatment on myopia control in children and adolescents, as compared to continuous treatment with orthokeratology, using a multicenter randomized controlled trial design. Subjects will be randomly assigned into either ortho-k and 0.01% atropine sequential treatment group or ortho-k continuous treatment group. Their axial length will be monitored over two years. Changes in axial length in the two groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 8-15 years old.
2. Spherical equivalent refractions (SERs) -0.50 to -6.00 Dioptres (D) and astigmatism less than -1.5 D in both eyes, anisometropia less than 1.5 D.
3. Best corrected visual acuity (BCVA) equal to or better than 20/25 in both eyes.
4. Bilateral intra-ocular pressure < 21mmHg.
5. Normal binocular and stereoscopic visual function.
6. Participants and their guardians' understanding and acceptance of random allocation of grouping.

Exclusion Criteria:

1. Manifest strabismus, except for intermittent tropia.
2. Ocular or systemic diseases which may affect vision or refractive error.
3. Previous use of myopia control without washout, including atropine, myopia control spectacles, myopia control contact lenses.
4. Other contraindications.

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 194 (Estimated)
Dates: Start 2024-09-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Axial length change | From baseline to the end of treatment at 25 months
  Axial length change (mm) is characterized as the difference between 25-month follow-up visit and baseline values. The IOLMaster or Lenstar are used to measure axial length (mm).

SECONDARY OUTCOMES:
Proportion of rapid myopia progression | From baseline to the end of treatment at 25 months
  Proportion of rapid myopia progression means the rate of cumulative axial growth ≥0.50 mm at 25 months) after intervention.
Axial length change | From baseline to 3, 6, 9, 12, and 19 months.
  Axial length change (mm) is characterized as the difference between 3, 6, 9, 12, and 19 months follow-up visit and baseline values. The IOLMaster or Lenstar are used to measure axial length (mm).
Incidence of adverse events | From baseline to 25 months.
  Incidence of adverse events is the rate of adverse events over the study period for subjects in both arms.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No